CLINICAL TRIAL: NCT03724825
Title: Correlation of Serum Adropin to Testosterone and Adiponectin in Obese Men
Status: Completed | Type: Observational
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Asmaa Abdel-mageed Muhammed, Assistant lecturer, Aswan University Hospital
Other Study IDs: Adropin in obese men
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Obesity; Dyslipidemias
Keywords: Adropin; adiponectin; testosterone; obese men
MeSH Terms: conditions — Obesity; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese men: Adult obese men (BMI ≥ 30 kg/m2)
  Interventions: Diagnostic Test: lipid profile: Total cholesterol (TC), triglycerides (TG), low density lipoprotein (LDL) and high density lipoprotein (HDL)); Diagnostic Test: Total testosterone; Diagnostic Test: Adropin; Diagnostic Test: Adiponectin
- normal men: normal weight men (18.5 ≤ BMI < 25 kg/m2 )
  Interventions: Diagnostic Test: lipid profile: Total cholesterol (TC), triglycerides (TG), low density lipoprotein (LDL) and high density lipoprotein (HDL)); Diagnostic Test: Total testosterone; Diagnostic Test: Adropin; Diagnostic Test: Adiponectin

INTERVENTIONS:
Diagnostic Test: lipid profile: Total cholesterol (TC), triglycerides (TG), low density lipoprotein (LDL) and high density lipoprotein (HDL)) — blood samples will be collected after 10 hours fasting
Diagnostic Test: Total testosterone — blood samples will be collected after 10 hours fasting
Diagnostic Test: Adropin — blood samples will be collected after 10 hours fasting
Diagnostic Test: Adiponectin — blood samples will be collected after 10 hours fasting

SUMMARY:
Obesity is associated with low testosterone in men and with dyslipidemia. Adropin hormone is negatively correlated with body mass index and is associated with dyslipidemia.

correlation between adropin and testosterone will be evaluated.

DETAILED DESCRIPTION:
Obesity, a worldwide epidemic is associated with multiple adverse health outcome as diabetes mellitus, hypertension and cardiovascular diseases caused mainly by dyslipidemia linked to obesity. Low testosterone levels in obese men were found associated with dyslipidemia.

Adropin is a new metabolic hormone that was first isolated in liver and brain tissues, It was observed that mice fed on a high-fat diet (HFD) had a rapid increase in adropin expression compared to control values. In human also, adropin levels were negatively correlated with body mass index (BMI) and were associated with dyslipidemia.

Adiponectin is a protein that is mainly produced by white adipose tissue and has an important role in lipid metabolism. Serum adiponectin concentrations were decreased in obese compared to normal weight men and significantly correlated with testosterone level.

ELIGIBILITY:
Inclusion Criteria:

Age from 18 years to 50 years. Clinically free except from obesity

Exclusion Criteria:

* Diabetes mellitus Hypertension Heart failure Kidney disease Smoking

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: obese and normal weight men from 18 years to 50 years
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
changes in lipid profile (TC, TG, LDL, HDL) levels | 6 months
  expected higher TC, TG, LDl levels and lower HDL levels in obese men compared to normal
changes in total testosterone levels | 6 months
  expected lower testosterone levels in obese men compared to normal men
changes in adropin level | 6 months
  expected lower adropin levels in obese men compared to normal men
changed in adiponectin levels | 6 months
  expected lower adiponectin level in obese men compared to normal men
correlation between adropin and testosterone | 6 months
correlation between adropin and adiponectin | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Abdelmageed Muhammed, Assistant lecturer, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University Hospital, Aswān, Egypt

REFERENCES:
- [Background] Canguven O, Talib RA, El Ansari W, Yassin DJ, Salman M, Al-Ansari A. Testosterone therapy has positive effects on anthropometric measures, metabolic syndrome components (obesity, lipid profile, Diabetes Mellitus control), blood indices, liver enzymes, and prostate health indicators in elderly hypogonadal men. Andrologia. 2017 Dec;49(10). doi: 10.1111/and.12768. Epub 2017 Mar 10. PMID 28295504
- [Background] Ghoshal S, Stevens JR, Billon C, Girardet C, Sitaula S, Leon AS, Rao DC, Skinner JS, Rankinen T, Bouchard C, Nunez MV, Stanhope KL, Howatt DA, Daugherty A, Zhang J, Schuelke M, Weiss EP, Coffey AR, Bennett BJ, Sethupathy P, Burris TP, Havel PJ, Butler AA. Adropin: An endocrine link between the biological clock and cholesterol homeostasis. Mol Metab. 2018 Feb;8:51-64. doi: 10.1016/j.molmet.2017.12.002. Epub 2017 Dec 30. PMID 29331507
- [Background] Yosaee S, Khodadost M, Esteghamati A, Speakman JR, Shidfar F, Nazari MN, Bitarafan V, Djafarian K. Metabolic Syndrome Patients Have Lower Levels of Adropin When Compared With Healthy Overweight/Obese and Lean Subjects. Am J Mens Health. 2017 Mar;11(2):426-434. doi: 10.1177/1557988316664074. Epub 2016 Aug 22. PMID 27550773
- [Background] Kim AY, Park YJ, Pan X, Shin KC, Kwak SH, Bassas AF, Sallam RM, Park KS, Alfadda AA, Xu A, Kim JB. Obesity-induced DNA hypermethylation of the adiponectin gene mediates insulin resistance. Nat Commun. 2015 Jul 3;6:7585. doi: 10.1038/ncomms8585. PMID 26139044
- [Background] Thomas S, Kratzsch D, Schaab M, Scholz M, Grunewald S, Thiery J, Paasch U, Kratzsch J. Seminal plasma adipokine levels are correlated with functional characteristics of spermatozoa. Fertil Steril. 2013 Apr;99(5):1256-1263.e3. doi: 10.1016/j.fertnstert.2012.12.022. Epub 2013 Jan 30. PMID 23375204
- [Derived] Muhammed AA, Eid RMHM, Mohammed WS, Abdel-Fadeil MR. An association between adropin hormone and total testosterone in obese men: a case-control study. BMC Endocr Disord. 2022 Jul 27;22(1):192. doi: 10.1186/s12902-022-01102-7. PMID 35897011